CLINICAL TRIAL: NCT05001672
Title: The Efficacy of TAF as a Prophylactic Antiviral Agent for HBsAg-positive Patients Receiving Biological DMARDs (bDMARDs)
Brief Title: The Efficacy of Prophylactic TAF for HBsAg-positive Patients Receiving bDMARDs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IN-TW-320-6150
Record Dates: First submitted 2021-07-02; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: HBV; Inflammatory Arthritis
MeSH Terms: conditions — Arthritis | interventions — tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Patients who fulfilled in all inclusion and exclusion criteria will be randomized into TAF 25mg qd or observation arm in 1:1 ratio.
  * 54 patients will be randomized into TAF arm*.
  * 54 patients will be randomized into observation arm initially.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAF arm (Experimental): 54 patients will be randomized into TAF arm*. TAF 25 mg QD will be initiated 7 days before bDMARDs, and continued for up to 144-weeks.
  *for patients received rituximab (anti-CD20 monoclonal antibody) will be enrolled into TAF arm, and TAF 25 mg QD will be initiated 7 days before rituximab, and continued for up to 144-weeks. Max 20 rituximab patients will be recruited.
  Interventions: Drug: Tenofovir alafenamide
- Observation arm (Other): 54 patients will be randomized into observation arm initially. These patients will be closely monitored their HBV status (including qHBsAg and HBV DNA) for 48 weeks. TAF 25 mg QD will be initiated for 144 weeks in the presence of HBV reactivation, or after 48 weeks of observation.
  Interventions: Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Tenofovir alafenamide — Tenofovir alafenamide (TAF, brand name: Vemlidy) is a hepatitis B virus nucleotide reverse transcriptase inhibitor oral medication for the treatment of chronic hepatitis B virus infection. It is a prodrug of tenofovir. Closely related to the commonly used reverse-transcriptase inhibitor tenofovir disoproxil fumarate, TAF has greater antiviral activity and better distribution into lymphoid tissues than that agent. Vemlidy was approved by the U.S. Food and Drug Administration (FDA) in November 2016 and the TAIWAN Food and Drug Administration (TFDA) in April 2017.
  Other Names: Vemlidy; TAF

SUMMARY:
Hepatitis B virus reactivation (HBVr) is an emerging issue and a potentially life-threatening complication to patients with history of Hepatitis B virus (HBV) infection whose immune system is deficient or suppressed. It is estimated that the risk of HBVr ranges 20%-50% in hepatitis B surface antigen (HBsAg)-positive patients undergoing chemotherapy or immunosuppressive therapy. Not only HBsAg-positive patients but also HBsAg-negative/antibody to hepatitis B core antigen (anti-HBc)-positive patients (resolved hepatitis B) have the risk of HBVr.

Recent studies also reported that the risk of HBVr associated with TNF-α inhibitor treatment widely ranged from 12.3% to 62.5%. Antiviral prophylaxis by nucleos(t)ide analogues (NUCs) is recommended for patients with high risk of HBVr according to 2018 AASLD guidance. Phase 3 studies reported that tenofovir alafenamide (Vemlidy, TAF) can effectively suppress HBV in both HBeAg-positive and HBeAg-negative chronic hepatitis B patients, and TAF is superior to TDF in safety profiles and ALT normalization. However, the evidence of TAF in prevention HBV reactivation for patients with HBsAg-positive and imflammatory arthritis, who need bDMARDs are still missing.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is the major cause of chronic hepatitis, liver cirrhosis and hepatocellular carcinoma. There are up to 248 million people worldwide chronically infected with HBV. HBV reactivation (HBVr) is an emerging issue and a potentially life-threatening complication to patients with history of HBV infection whose immune system is deficient or suppressed. It is estimated that the risk of HBVr ranges 20%-50% in hepatitis B surface antigen (HBsAg)-positive patients undergoing chemotherapy or immunosuppressive therapy. Not only HBsAg-positive patients but also HBsAg-negative/antibody to hepatitis B core antigen (anti-HBc)-positive patients (resolved hepatitis B) have the risk of HBVr. The investigator's studies have demonstrated that the risk of HBsAg seroreversion was 10% in diffuse large B cell lymphoma patients undergoing anti-CD20 (rituximab) treatment; and the risk of HBsAg reverse seroconversion in rheumatic arthritis (RA) patients with resolved HBV infection and received biological disease-modifying antirheumatic drugs (bDMARDs) or glucocorticoid (GC) treatment can persist for up to 10 years. In the investigator's previous study, it also be investigated the risk of HBVr under different immunosuppressant regimens in HBsAg-positive patients with RA, and the investigator pointed out immunosuppressive treatment with a combination of GC, synthetic disease-modifying antirheumatic drugs (sDMARDs), and bDMARDs has the highest risk of HBVr with annual incidence around 20%. Recent studies also reported that the risk of HBVr associated with TNF-α inhibitor treatment widely ranged from 12.3% to 62.5%.

Antiviral prophylaxis by nucleos(t)ide analogues (NUCs) is recommended for patients with high risk of HBVr according to 2018 AASLD guidance. Phase 3 studies reported that tenofovir alafenamide (Vemlidy, TAF) can effectively suppress HBV in both HBeAg-positive and HBeAg-negative chronic hepatitis B patients, and TAF is superior to TDF in safety profiles and ALT normalization. However, the evidence of TAF in prevention HBV reactivation for patients with HBsAg-positive and imflammatory arthritis, who need bDMARDs are still missing. Therefore, the investigator plans to conduct this randomized controlled trial to confirm the efficacy of TAF as a prophylactic antiviral agent for HBsAg-positive patients with inflammatory arthritis (IA) on bDMARDs treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >=20 years old;
* History of chronic hepatitis B with HBsAg-positive;
* Both HBeAg-positive and HBeAg-negative are allowed;
* Inflammatory arthritis (including psoriatic arthritis);
* On bDMARDs treatment or will start bDMARDs within in 4 weeks. The bDMARDs included all anti-TNF-α agents, rituximab (anti-CD20 monoclonal antibody), tocilizumab (anti-interleukin 6 receptor monoclonal antibody), abatacept (cytotoxic T-lymphocyte-associated antigen 4 immunoglobulin), and all new biologics with indication of IA treatment;
* No NUCs treatment in recent 6 months;
* No limitation of the baseline HBV DNA level;
* Total bilirubin level <2 mg/dL;
* ALT < 2x ULN (<80 U/L).

Exclusion Criteria:

* Child-Pugh class >B7;
* Active EV bleeding within 4 weeks;
* History of hepatic encephalopathy or intractable ascites;
* Coexist with other primary liver diseases, such as active chronic hepatitis C, hepatitis D, autoimmune hepatitis, or Wilson's disease. (*HCV RNA undetectable is allowed to enroll);
* Active malignancy;
* Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year HBV reactivation rate | Up to 1-year
  The assessment for the HBV reactivation is by the marker as hepatitis b viral load (unit: IU/ML).

SECONDARY OUTCOMES:
Serial change of renal and liver function | Up to 3-years
  The assessment for the renal function is by the markers as serum creatinine (unit: mg/dL), eGFR (unit: 60 mL/min/1.73M^2) and serum inorganic phosphorus (unit: mg/dL); for the liver function is by the markers as ALT/AST (unit: U/L) and child-pugh score.
  The child-pugh score is determined by scoring five clinical measures of liver disease. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe, and the five clinical measures are: total bilirubin (unit: mg/dL), serum albumin (unit: g/dL), prothrombin time (unit: sec), absence/presence of ascites and absence/presence of hepatic encephalopathy. The higher scores mean a worse outcome.
Observation of bone mineral density at 48-weeks, 96-weeks, and 144-weeks | Up to 3-years
  The assessment for the bone mineral density is by the marker as T-score.
The 1-year virological remission rate | Up to 1-year
  The assessment for the HBV reactivation is by the marker as hepatitis b viral load (unit: IU/ML).
The 1-year HBeAg seroconversion rate | Up to 1-year
  The assessment for the HBeAg seroconversion is by the marker as HBeAg (unit: COI).
The adverse reactions and compliance | Up to 3-years
  The assessment for the adverse reactions is by the CTCAE v5.0, and the compliance is by the residual study drug.

IPD SHARING:
Plan to Share IPD: No